CLINICAL TRIAL: NCT00941681
Title: An Open Label Study to Investigate the Pharmacokinetics of CK-1827452 Administered Orally to Patients With Stable Heart Failure
Brief Title: Pharmacokinetics of Oral CK-1827452 in Patients With Stable Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CY 1021
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Heart Failure
Keywords: omecamtiv mecarbil
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: MR 50 mg BID (Experimental): Modified-release (MR) 50 mg dose of CK-1827452 twice a day (BID) for 10 days.
  Interventions: Drug: CK-1827452
- Cohort 2: IR 37.5 mg TID (Experimental): Immediate-release (IR) 37.5 mg dose of CK-1827452 three times a day (TID) for 10 days.
  Interventions: Drug: CK-1827452
- Cohort 3: MR 100 mg BID (Experimental): Modified-release (MR) 100 mg dose of CK-1827452 twice a day (BID) for 10 days
  Interventions: Drug: CK-1827452

INTERVENTIONS:
Drug: CK-1827452 — 50 mg MR CK-1827452 BID for 10 days
  Arms: Cohort 1: MR 50 mg BID
Drug: CK-1827452 — 37.5 mg IR CK-1827452 TID for 10 days
  Arms: Cohort 2: IR 37.5 mg TID
Drug: CK-1827452 — 100 mg MR CK-1827452 BID for 10 days
  Arms: Cohort 3: MR 100 mg BID

SUMMARY:
This study is designed to understand the pharmacokinetics of different oral formulations of CK-1827452 being considered for future studies in patients with heart failure. This study will compare the pharmacokinetics and safety and tolerability of both modified-release (MR) and immediate-release (IR) oral formulations of CK-1827452.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed an Informed Consent Form/Patient Information Sheet for this study approved by the governing Institutional Review Board (IRB) or Independent Ethics Committee (IEC)
2. The patient is at least 18 years old at the time of consent
3. Left ventricular ejection fraction (LVEF) ≤ 35% as determined by the Investigator within 3 weeks prior to enrollment
4. Treated for at least 4 weeks with a beta blocker and an ACE inhibitor (and/or an ARB) unless not tolerated. If prescribed, diuretics must have been administered according to a consistent regimen for at least 4 weeks.
5. Diagnosed with heart failure for ≥ 3 months prior to enrollment
6. Patient is considered to be an appropriate candidate for study enrollment as determined by the patient's clinical laboratory findings, vital signs and ECGs within normal range, or if outside of the normal range not deemed clinically significant in the opinion of the Investigator
7. For female patients only: The patient is post-menopausal (≥ 1 year) or sterilized, or if she is of childbearing potential, she is not breastfeeding, her pregnancy test is negative, she has no intention to become pregnant during the course of the study, and she is using contraceptive drugs or devices. For male patients only: Male patients agree for the duration of the study and 10 weeks after the end of the study to use a condom during sexual intercourse with female partners who are of reproductive potential and to have female partners use an additional effective means of contraception (eg, diaphragm plus spermicide, or oral contraceptives) or the male subject must agree to abstain from sexual intercourse for 10 weeks after the end of the study.

Exclusion Criteria:

1. Patient has been hospitalised for heart failure, acute coronary syndrome, myocardial infarction, coronary revascularisation, transient ischemic attack or stroke, cardiac arrhythmia, or major surgery within 6 weeks prior to enrollment
2. Poorly controlled hypertension defined as blood pressure > 150/95 mmHg, documented on at least 2 separate occasions prior to enrollment
3. The patient has a supine heart rate ≥ 100 beats per minute after 10 minutes of rest
4. Patient has a troponin I at screening that is above the upper limit of normal
5. The patient has severe aortic or mitral stenosis
6. The patient has active myocarditis; clinically significant restrictive, constrictive, or hypertrophic obstructive cardiomyopathy; clinically significant congenital heart disease; history of major organ transplantation
7. The patient has Canadian Cardiovascular Society Class IV angina
8. Patient is on chronic anti-arrhythmic therapy, with the exception of amiodarone
9. Patient has impaired renal function defined as an estimated GFR ≤ 30 ml/min/1.73 m2 calculated by the Modification of Diet in Renal Disease (MDRD) equation
10. Patient is currently taking, or has taken within 14 days prior to enrollment, a potent CYP3A4 inhibitor (medication or food). Patient is currently taking, or has taken within 28 days prior to enrollment, a potent CYP3A4 inducer (medication or food).
11. The patient has hepatic impairment defined as a total bilirubin > 3 mg/dL, or an ALT or AST > 2 times the upper limit of normal
12. Concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 1 year
13. The patient has received an investigational drug or device within 30 days or 5 half-lives, whichever is greater, of enrollment
14. Patient has, in the opinion of the Investigator, a condition that compromises the ability of the subject to give written informed consent or to comply with study procedures, including scheduled self-administration of oral CK-1827452
15. The patient has had any prior treatment with CK-1827452

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Georgia (3):
  - Cardio-Reanimation Centre, Tbilisi
  - Diagnostic Services Clinic, Tbilisi
  - Tbilisi State Medical University Clinic #1, Tbilisi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Started | 12 | 11 | 12
Completed | 12 | 10 | 12
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID | Total
Number analyzed (Participants) | 12 | 11 | 12 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 6 | 21
  >=65 years | 5 | 3 | 6 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.74) | 61.1 (7.97) | 62.4 (11.51) | 62.6 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 11
  Male | 8 | 8 | 8 | 24
Region of Enrollment [Number; unit: participants]
  Georgia | 12 | 11 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: C Max (Day 1, Dose 1)
Description: Maximum plasma concentration (C max) measured in nanograms per milliliter (ng/mL) post first dose and pre second dose on day 1. Doses are approximately 12 hours apart in cohort 1 and 3 and 8 hours apart in cohort 2.
Time Frame: 1 day
Population: PK population (4 patients excluded from cohort 3 analysis due to improper dosing).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Number analyzed (Participants) | 12 | 11 | 8
ng/mL | 58 (27) | 243 (148) | 209 (164)

2. Secondary Outcome: Evaluate the Safety and Tolerability of Oral Formulations of CK-1827452 When Dosed to Steady-state in Patients With Stable Heart Failure.
Time Frame: 1 week
Reporting Status: Not Posted

3. Primary Outcome: T Max (Day 1, Dose 1)
Description: Time of observed maximum plasma concentration (T max) measured in hours (hr) post first dose and pre second dose on day 1. Doses are approximately 12 hours apart in cohort 1 and 3 and 8 hours apart in cohort 2.
Time Frame: 1 day
Population: PK population (4 patients excluded from cohort 3 analysis due to improper dosing).
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Number analyzed (Participants) | 12 | 11 | 8
hr | 3.5 (2.9) | 3.7 (3.7) | 3.5 (3.9)

4. Primary Outcome: AUC (Day 1, Dose 1)
Description: Area under the curve (AUC) measured in hours * nanograms per milliliter (hr*ng/mL) post first dose and pre second dose on day 1. Doses are approximately 12 hours apart in cohort 1 and 3 and 8 hours apart in cohort 2.
Time Frame: 1 day
Population: PK population (4 patients excluded from cohort 3 analysis due to improper dosing).
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Number analyzed (Participants) | 12 | 11 | 8
hr*ng/mL | 446 (206) | 1003 (387) | 1650 (1354)

5. Primary Outcome: C Max (Day 10)
Description: Maximum plasma concentration (C max) measured in nanograms per milliliter (ng/mL) post dose on day 10. Only one dose was administered on day 10 (final dose of study).
Time Frame: 1 day
Population: PK population (4 patients excluded from cohort 3 analysis due to improper dosing and 1 patient excluded from cohort 2 due to sudden death).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Number analyzed (Participants) | 12 | 10 | 8
ng/mL | 205 (111) | 420 (158) | 704 (494)

6. Primary Outcome: T Max (Day 10)
Description: Time of observed maximum plasma concentration (T max) measured in hours (hr) post dose on day 10. Only one dose was administered on day 10 (final dose of study).
Time Frame: 1 day
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Number analyzed (Participants) | 12 | 10 | 8
hr | 1.8 (0.9) | 1.8 (1.1) | 2.7 (1.6)

7. Primary Outcome: AUC (Day 10)
Description: Area under the curve (AUC) measured in hours * nanograms per milliliter (hr*ng/mL) post dose on day 10. Only one dose was administered on day 10 (final dose of study).
Time Frame: 1 day
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Number analyzed (Participants) | 12 | 10 | 8
hr*ng/mL | 1886 (1002) | 2118 (623) | 6457 (5147)

ADVERSE EVENTS:
Arm/Group | Cohort 1: MR 50 mg BID | Cohort 2: IR 37.5 mg TID | Cohort 3: MR 100 mg BID
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MR 50 mg BID (N=12) | Cohort 2: IR 37.5 mg TID (N=11) | Cohort 3: MR 100 mg BID (N=12)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) — Reported as unrelated to treatment by Investigator.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MR 50 mg BID (N=12) | Cohort 2: IR 37.5 mg TID (N=11) | Cohort 3: MR 100 mg BID (N=12)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to publish the results of the trial in collaboration with the Investigators.